CLINICAL TRIAL: NCT05663632
Title: Triglyceride-Glucose Index In Heart Failure Patients In Sohag University Hospital
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Aliaa Khairy Shabaan, resident at internal medicine department, Sohag University
Other Study IDs: Soh-Med-22-12-04
Record Dates: First submitted 2022-12-15; First posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Heart Failure; Insulin Resistance
Keywords: heart failure; triglyceride-glucose index
MeSH Terms: conditions — Heart Failure; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group 1 heart failure patients
- Group 2 controle

SUMMARY:
study the relationship between Triglyceride glucose index and heart failure patients

ELIGIBILITY:
Inclusion Criteria:

* All Heart Failure patients attend to sohag university hospital aged above 18 year old .

Exclusion Criteria:

* Patients on lipid lowering medications
* Patients on antidiabetic drugs
* Patients with comorbidities eg liver cirrhosis or malignancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be divided into2 groups, as following:
  Group (1) Heart Failure patients (100 patients) Group (2) control group(100 person)
  All groups will be subjected to :
  1. Complete history taking with special emphasis on Age ,Sex, Smoking, Diabetes mellitus and Hypertension.
  2. A thorough clinical examination will stress on:
  1- Heart rate (b.p.m.). 2-Systolic BP (mmHg). 3-BMI calculated as the ( weight (kg)/height (m)2). 3-The following investigations will be done to every subject:
  1. FBG (mg/dL)
  2. FTG, (mg/dL)
  3. Total cholesterol (TC) (mg/dL)
  4. SCr (mg/dL)
  5. Echocardiography
  TyG index is calculated as ln [fasting triglyceride (mg/dL) * fasting glucose (mg/dL) / 2]
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Triglyceride-Glucose Index in Heart Failure Patients | 6 months
  identify the relationship between Triglyceride-Glucose Index and heart failure patients in Sohag University hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

REFERENCES:
- [Background] GBD 2019 Diseases and Injuries Collaborators. Global burden of 369 diseases and injuries in 204 countries and territories, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet. 2020 Oct 17;396(10258):1204-1222. doi: 10.1016/S0140-6736(20)30925-9. PMID 33069326
- [Background] Davison B, Cotter G. Why is heart failure so important in the 21st century? Eur J Heart Fail. 2015 Feb;17(2):122-4. doi: 10.1002/ejhf.219. Epub 2014 Dec 30. No abstract available. PMID 25557121
- [Background] Miller M, Seidler A, Moalemi A, Pearson TA. Normal triglyceride levels and coronary artery disease events: the Baltimore Coronary Observational Long-Term Study. J Am Coll Cardiol. 1998 May;31(6):1252-7. doi: 10.1016/s0735-1097(98)00083-7. PMID 9581716
- [Background] Shaye K, Amir T, Shlomo S, Yechezkel S. Fasting glucose levels within the high normal range predict cardiovascular outcome. Am Heart J. 2012 Jul;164(1):111-6. doi: 10.1016/j.ahj.2012.03.023. PMID 22795290